CLINICAL TRIAL: NCT06906601
Title: Preoperative Magnetic Tracking in Breast Surgery in France: French Medical-economic Study.
Acronym: MAGNETO
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET24-213 (MAGNETO)
Record Dates: First submitted 2025-03-18; First posted 2025-04-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Medico-economic Impact; Breast Cancer Surgery
Keywords: cancer; breast cancer; breast cancer surgery; preoperative localization; magnetic clip; wire localization; health economic study; Cost-consequence analysis; medico-economic
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- magnetic clip localization: The preoperative localization can be performed using several techniques, magnetic clip localization will be use in this cohort
  Interventions: Procedure: magnetic clip localization; Procedure: Breast cancer surgery
- wire localization: The preoperative localization can be performed using several techniques, wire localization will be use in this cohort
  Interventions: Procedure: metallic wire localization.; Procedure: Breast cancer surgery

INTERVENTIONS:
Procedure: magnetic clip localization — magnetic clip localization for preoperative localization for breast cancer surgery
  Groups: magnetic clip localization
Procedure: metallic wire localization. — metallic wire localization for preoperative localization for breast cancer surgery
  Groups: wire localization
Procedure: Breast cancer surgery — Patient with invasive or in situ breast carcinoma, presenting with a unifocal and unilateral lesion, requiring a first-line breast-conserving treatment with preoperative localization, regardless of the associated lymph node procedure

SUMMARY:
MAGNETO is a French medico-economic study on preoperative localization in breast cancer surgery. The main objective is to conduct a cost-consequence analysis comparing magnetic clip localization with the use of metallic wires for the preoperative identification of non-palpable breast lesions. The choice of localization method is left to the physician's and center's discretion. The study is non-interventional (with only questionnaires and data collection), prospective, and multicenter, with patient follow-up lasting up to six months after breast surgery.

DETAILED DESCRIPTION:
The MAGNETO study is a non-interventional, prospective, and multicenter study. It includes two cohorts: one using magnetic clip localization and the other using metallic wire localization.

Patients are enrolled by the surgeon during the preoperative consultation validating the conservative surgery with preoperative localization. The choice of cohort is left to the discretion of the center based on their routine practice. Baseline data, including patient and disease characteristics, are collected.

Depending on the assigned cohort, localization is performed either with a magnetic clip or a metallic wire. A mammogram is then performed to assess the correct positioning of the marker and its distance from the target lesion. At this stage, the radiologist completes a Likert scale satisfaction questionnaire.

Breast-conserving surgery is performed according to the hospital's standard practices. On the day of the procedure, the surgeon also completes a Likert scale satisfaction questionnaire.

Patients complete quality of life (EQ-5D-5L) and satisfaction questionnaires at several points throughout the study. Postoperative complications are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* I1. Female aged ≥ 18 years;
* I2. Patient presenting with a unifocal and unilateral lesion of invasive carcinoma or in situ;
* I3. Indication for first breast-conserving treatment with the need for preoperative localization of the lesion, regardless of the associated lymph node procedure;
* I4. Patient affiliated with a health insurance system;
* I5. Non-opposition to the study.

Exclusion Criteria:

* E.1. Psychological, family, or sociological condition that may potentially compromise adherence to the treatment protocol and follow-up;
* E.2. Bilateral surgery required;
* E.3. Patient with metastatic breast cancer;
* E.4. Multifocal or benign lesions;
* E.5. Pregnant or breastfeeding patient;
* E.6. Need for neoadjuvant treatment;
* E.7. Associated breast reduction procedure;
* E.8. Patient under guardianship, curatorship, or deprived of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cisgender female with breast cancer
Study Population: Patients recruited in 9 centers spread across France
Sampling Method: Non-Probability Sample
Enrollment: 772 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of the average total cost of patient care with magnetic clip localization versus the use of a hookwire, up to 6 months post-surgery | 6 months post surgery
  Effectiveness of localization in terms of lesion identification (did the localization, based on the pathological report, allow the lesion to be located in the breast?)
  * Rate of clear margins (for isolated in situ lesions: margin ≥ 2 mm, and for invasive cancers: non-zero margin)
  * Percentage of patients requiring re-intervention due to an unclear margin
  * Measured distance between the marker and the target lesion during the procedure
  * Ratio between the weight of the resected specimen and the lesion size in g/mm²
  * Patient satisfaction with their care, assessed using a 5-point Likert scale during the postoperative consultation (between day 15 and day 30 after resection)
  * Radiologist satisfaction with the marker placement, assessed using a 5-point Likert scale immediately after placement
  * Surgeon satisfaction with lesion localization, assessed using a 5-point Likert scale at the end of the surgery.

SECONDARY OUTCOMES:
Quality of life of patientes | At inclusion, 15 to 30 days after surgery and 6 months after surgery
  Quality of life assessed using the 5-level EQ-5D version (EQ-5D-5L).The questionnaire assesses 5 dimensions (Mobility, Self-care, Usual activities, Pain/Discomfort, Anxiety/Depression). Each dimension is rated on 5 levels (from 1 = no problems to 5 = extreme problems).
Satisfaction of radiologist and surgeon | Within 24 hours after the maker placement and within 24 hours after the surgery
  Questionnaire to evaluate the satisfaction of radiologist after the maker placement and questionnaire to evaluate the satisfaction of surgeon after the surgery. The score isn't on a scale.
Patient satisfaction and experience. | 15 to 30 days after surgery
  Questionnaire after the surgery to evaluated the patient satisfaction and experience. The score isn't on a scale.
Budget impact analysis of pre operative magnetic clip localization versus the use of a hookwire. | At 1, 2 and 3 years
  The decision to include a Budget Impact Analysis (BIA) in this study is in line with the framework agreement signed in January 2016 between the Economic Committee for Medicinal Products (Comité Economique des Produits de Santé - CEPS, in French) and the Pharmaceutical Industry (Les Entreprises du Médicament - LEEM, in French), which advises the implementation of a BIA in addition to the medico-economic study. The BIA will strictly comply with the HAS requirements presented in its methodological guide for BIA.
  A budget impact model (BIM) will be developed with the French National health insurance perspective. The cost of the current (hookwire) or new intervention (magnetic clip) mix will be assessed. The population to be included in a BIA will be all patients eligible in France for the new intervention during the time horizon of 3 years. The results will be expressed in incremental budget impact in the first, second and third year.
The organisationnal impact of magnetic clip versus metallic wires. | At 6 months
  The organizational analysis will be based on performance indicators of magnetic clips compared to metallic wires, such as the number of patient visits to the hospital before surgery, the number of localization procedures performed on the day of the intervention, the length of stay, waiting times, and the number of emergency visits throughout the follow-up period. The stochastic variables (lengths of stay, intervals between stays) will be modeled using appropriate statistical distributions, determined by maximum likelihood estimation based on statistical analyses of the extracted data.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hospices Civils de Lyon Hopital de la Croix rousse, Lyon
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Lorraine (ICL), Nancy
  - Hôpital Nord -Ouest Val d'Oise (NOVO), Pontoise
  - Institut GODINOT, Reims
  - Institut de Cancérologie de l'Ouest Rene Gauducheau, Saint-Herblain
  - IUCT-Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif